CLINICAL TRIAL: NCT05163678
Title: Evaluation of the Future of Adolescents and Young Adults Received in an Early Care System
Acronym: ReFSEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Santé des Étudiants de France (Other)
Responsible Party: Sponsor
Other Study IDs: FSEF
Record Dates: First submitted 2021-11-17; First posted 2021-12-20 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-11

CONDITIONS: Psychological Distress
Keywords: psychic; early treatment; Adolescent and young adults; cohort follow up; epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient group: All adolescents or young adults presenting for a consultation in the FSEF "Relais" systems.
  They will be assessed upon entry into the device (T0), at the end of the follow-up (T1) and 6 months after the end of the follow-up (T6).
  Interventions: Other: monitoring naturalistic of cohort

INTERVENTIONS:
Other: monitoring naturalistic of cohort — Assessment at the start of care in the "Relais" (T0), at the end (T1) and 6 months later (T6).

SUMMARY:
This is a prospective clinical epidemiology study based on the naturalistic follow-up of a cohort of 1 500 young people aged 11 to 25 presenting consecutively over the course of one year at the Relais d'Ile de France.

Young people will be assessed on entry into the system (T0), at the end of the follow-up (T1) and 6 months after the end of the follow-up (T6).

DETAILED DESCRIPTION:
Psychic suffering is very common among young people; a public health issue in France is to improve its early identification and treatment. To this end, the Fondation Santé des Etudiants de France (FSEF) has developed ambulatory systems in France called "Relais Collégiens-Lycéens-Etudiants" offering adolescents and young adults a reception, evaluation and support or a quick referral.

The FSEF Relay system allows a wide range of subjects to benefit from rapid support for a situation of mental suffering, which specialized care structures cannot do. In fact, first of all, if the school teams and the entourage are not made aware of the need to be attentive to psychological suffering, it is not detected, then when it is, most of these young people are not. not addressed out of reluctance from those around them or from the young person himself who refuse to go to psychiatric care experienced as stigmatizing; then, when young people are referred to care structures, consultation times are unsuitable (saturated structures) while these young people need a rapid response. The impact of early detection systems in adolescence has been little studied, this research proposes to initiate such an approach on a large panel of young people from a systematic evaluation, by evaluating the future in the short and medium term.

This research proposes to assess the impact of these devices. T his is a prospective clinical epidemiology study based on the naturalistic follow-up of a cohort of 1,500 young people aged 11 to 25 presenting consecutively over the course of one year at the 5 Relais d'Ile de France. Young people will be assessed on entry into the system (T0), at the end of the follow-up (T1) and 6 months after the end of the follow-up (T6). The data collected will be:

* The state of health (including mental health, somatic health and drug consumption), lifestyle and education and social adaptation through clinical assessment and self-questionnaires completed by young people:
* The clinical assessment includes the following elements: the severity of the psychological suffering (CGI, Global Clinical Impression), the psychosocial impact (SOFAS, Social and Occupational Functioning Assessment Scale) and the diagnosis of mental disorder according to the ICD 10 (International Classification) 10th Revision) when relevant.
* The self-questionnaires assess psychological suffering (K10, Kessler scale 10 items), social functioning (WSAS, Work Social Adjustment Scale) as well as satisfaction with the care provided (CSQ-8, Client Satisfaction Questionnaire 8 items, and Likert scale, at T1 and T6).
* The EDGAR grid (Interview, Approach, Group, Support, Meeting) to quantify the care offered at the Relais and their cost.
* The orientation that may be offered following this support

ELIGIBILITY:
Inclusion Criteria:

* All adolescents, young adults in the age group 11-25 years,
* Presenting ill-being or psychological suffering, living in the health area concerned,
* Arriving alone or accompagniead at the "Realis" during the sudy period
* Agreeing to participate.

Exclusion Criteria:

* Young people outside the 11-25 age group,
* Parents and children who do not speak French or who cannot read or write.
* Young people in crisis situations requiring immediate hospitalization without consultation at the Relais.
* Refusal to participate

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will focus on 1500 files of young people aged 11 to 25, received in consultation in the Relays over one year (average activity in recent years). Participation will be voluntary.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Detailed description of the socio-demographic characteristics of the population hosted in the Relais | To the inclusion of young people
  Socio-demographic description of the population (Sex, age,nationality, civil and family situation, education)
Detailed description of the socio-demographic characteristics of the population hosted in the Relais | To the inclusion of young people
  By whom it is addressed, the reasons for addressing it, the level of mental suffering, the severity of the situation (diagnostic).
Detailed description of the socio-demographic characteristics of the population hosted in the Relais | To the inclusion of young people
  The psycho-social impact of the difficulties will also be assessed, also including data on the school career and the types and intensity of care generated, the duration of the follow-up, the diagnosis made and the orientation proposed, if applicable.

SECONDARY OUTCOMES:
The futur of young people taken care of in the "Relais" | End of care (care between 6 months to 1 year) and 6 months after end of follow-up
  Assessment of the fate at the end of the care and at 6 months, of adolescents and young adults received at least once as part of a consultation in a Relay. The criteria will relate to the assessment at the end of treatment and then at 6 months there of, in comparison with the initial state. These comparisons will relate to the level of psychological suffering, the psycho-social impact, and the implementation of the recommended care.
Satisfaction of subjects and his parents | End of care (care between 6 months to 1 year) and 6 months after end of follow-up
  Evaluate the level of satisfaction by means of a questionnaire of the subject and his parents with regard to the intervention and the orientation within the framework of the Relay schemes at the end of the care and at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Godart, PU-PH, Principal Investigator — Fondation Santé des Étudiants de France
Locations (3):
- France (3):
  - Relais - Centre Adour, Aire-sur-l'Adour
  - Relais 77, Neufmoutiers-en-Brie
  - Relais 93 - Sceaux, Sceaux

IPD SHARING:
Plan to Share IPD: No